CLINICAL TRIAL: NCT06819345
Title: Patients and Health Providers Experience and Choice of Treatment in End Stage Renal Disease
Brief Title: Impact of PREMs in the Shared Decision Process for Renal Replacement Treatment Methods.
Acronym: PEACE
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 908
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease, Stage 4 (Severe); Chronic Kidney Disease, Stage 5
Keywords: Chronic kidney disease; renal replacement therapy,; caregivers; PREM; PROM; shared decision making
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: -Patients with chronic renal disease stage 4-5 not on dialysis followed by a nephrologist for at least three months.
  Interventions: Other: Survey form
- Caregivers: First non-professional natural caregiver identified by the patient for all voluntary caregivers.
  - Caregiver with a sufficient level of oral comprehension of French, able to understand the research
  Interventions: Other: Survey form
- Health professionals: Nephrologists and nurses or other health professionals caring for patients included in the study.
  Interventions: Other: Survey form

INTERVENTIONS:
Other: Survey form — PPE15 (Picker Patient Experience Questionnaire) at all visit of the study KDQOL-SF (Kidney Disease Quality Of Life -short form) at inclusion and 3 months after initiation of RRT ou 24 months after inclusion SDMQ9 (Shared Decision Making Questionnaire): at inclusion and 3 months after receiving information related to RRT SDRS (Score Decision Regret Scale) : 3 months after initiation of RRT ou 24 months after inclusion HLS EU 16 (Health Literacy Survey) : at inclusion or 3 months after information on RRT

SUMMARY:
The French "my health 2022" plan is the first bundled payment initiative for stage 4 and 5 chronic kidney disease (CKD) pathway with the aim to improve the quality of care and promote a multi professional collaboration for a more holistic approach of healthcare. Renal Replacement therapies (RRT) have a significant impact on the quality of life and autonomy of patients and their caregivers. The transition to these treatments is a critical point in the pathway, involving a complex choice for patients that cannot be based solely on medical considerations but requires to assess the needs and preferences of patients and their caregivers in order to improve their experience and the quality of care. The investigators propose to conduct a prospective cohort study aimed at 1/ describing the patient and caregiver experience, patient related outcome measures (PROM) and the quality of life in relation to the decision-making process 2/ identifying the individual factors (socio-cultural, health literacy) associated with the patient experience, 3/ assessing the expectations and needs of patients regarding the information and support received during the process, and 4/ describing the perceptions of caregivers and professionals regarding the information provided and the decision-making process. The assessments will be conducted by questionnaires before, 3 months after the information on RRT and 3 months after the initiation of RRT or 24 months after the initial information for patients and caregivers and at the time of information on RRT for professionals. The data from the questionnaires will be further explored by a qualitative survey in a subgroup of patients and caregivers. The results of this study will help identify the factors determining the choice and satisfaction of patients and their caregivers in order to adapt the decision making support and thus have a patient-centered approach.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Stage 4-5 chronic kidney disease not on dialysis with a nephrologist follow up >3 months
* Glomerular filtration rate estimated by the CKD EPI formula < 20 ml/min/1.73 m2,
* Referred for consultation and information on renal replacement therapies.
* Age >18 years old.
* Patient with a sufficient level of oral comprehension of French, able to understand the research

Exclusion Criteria:

* significant cognitive disorders preventing decision making
* patients under guardianship, or legal protection
* referred for ultrafiltration in the context of cardio renal syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the CKD patients cohort followed at the nephrology department Hôpital Edouard Herriot with at least 3 months of follow up at the department and referred to the consultation for renal replacement therapies information.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient related experience measure (PREM) | 3 months after the announcement of stage V renal failure during the usual follow-up nephrology consultation And 3 months after the start of renal replacement therapy
  The main objective is to describe and monitor the evolution of the chronic renal failure patient experience during the decision-making process regarding renal replacement therapies (PD, HD or transplantation).
  Using the questionnaire : Picker Patient Experience PPE15

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology, Hypertension, dialysis department of Edouard Herriot hospital, Lyon, France